CLINICAL TRIAL: NCT02113748
Title: Downhill Walking to Enhance Training Effects in Patients With COPD
Brief Title: Downhill Walking Training in COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: Research Foundation Flanders (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Thierry Troosters, Prof., KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML10278
Record Dates: First submitted 2014-04-08; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary disease, chronic obstructive; Downhill walking; exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Downhill walking training (Experimental): Exercise training including treadmill walking with a negative inclination.
  Interventions: Other: Downhill walking training
- Conventional walking training (Active Comparator): Exercise training including treadmill walking without inclination. Possible to progress training intensity with positive inclinations.
  Interventions: Other: Conventional walking training

INTERVENTIONS:
Other: Downhill walking training — Walk on a treadmill with a negative inclination.
  Arms: Downhill walking training
Other: Conventional walking training — Walk on a treadmill without inclination. Possible to progress training intensity with positive inclinations
  Arms: Conventional walking training

SUMMARY:
This randomized control trial will investigate whether a modality that generates more contractile muscle fatigue with lower ventilatory requirements render better results after a 12-week exercise training program in subjects with COPD.

Subjects will be randomized to either exercise in a training program including downhill walking or to exercise in a training program including conventional walking.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of COPD according to internationally accepted guidelines
* Patients referred to the outpatient PR program of Gasthuisberg University Hospital(Leuven, Belgium)

Exclusion Criteria:

* Any underlying disease or musculoskeletal limitation that could impair the ability to perform any of the exercise training modalities
* Absence of exacerbations in the previous month before entering the present study
* Patients included on the waiting list for lung transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
changes in 6-minute walking distance | changes from baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Troosters, PhD, Principal Investigator — KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vl-Brabant, Belgium

REFERENCES:
- [Derived] Camillo CA, Osadnik CR, Burtin C, Everaerts S, Hornikx M, Demeyer H, Loeckx M, Rodrigues FM, Maes K, Gayan-Ramirez G, Janssens W, Troosters T. Effects of downhill walking in pulmonary rehabilitation for patients with COPD: a randomised controlled trial. Eur Respir J. 2020 Sep 17;56(3):2000639. doi: 10.1183/13993003.00639-2020. Print 2020 Sep. PMID 32444407